CLINICAL TRIAL: NCT03675880
Title: A Phase Ⅰ Clinical Study of TAB014 in Wet( Neovascular)Age-related Macular Degeneration(AMD) Subjects
Brief Title: TAB014(Drug Code) in Wet( Neovascular)Age-related Macular Degeneration(AMD) Subjects
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lee's Pharmaceutical Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZK-TAB-201709
Record Dates: First submitted 2018-09-05; First posted 2018-09-18 (Actual); Last update posted 2018-09-26 (Actual); Status verified 2018-09

CONDITIONS: AMD

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- 1.25mg(0.05ml) single-dose (Experimental): Eight subjects will be treated with TAB014 1.25mg(0.05ml) single-dose
  Interventions: Drug: TAB014
- 2.00mg(0.08ml) single-dose (Experimental): Eight subjects will be treated with TAB014 2.00mg(0.08ml) single-dose
  Interventions: Drug: TAB014
- 2.50mg(0.10ml) single-dose (Experimental): Eight subjects will be treated with TAB014 2.50mg(0.10ml) single-dose
  Interventions: Drug: TAB014
- 1.25mg(0.05ml) multiple-dose (Experimental): Eight subjects will be treated with TAB014 1.25mg(0.05ml) multiple-dose after 1.25mg(0.05ml) single-dose
  Interventions: Drug: TAB014
- 2.00mg(0.08ml) multiple-dose (Experimental): Eight subjects will be treated with TAB014 2.00mg(0.08ml) multiple-dose after 2.00mg(0.08ml) single-dose
  Interventions: Drug: TAB014
- 2.50mg(0.10ml) multiple-dose (Experimental): Eight subjects will be treated with TAB014 2.50mg(0.10ml) multiple-dose after 2.50mg(0.10ml) single-dose
  Interventions: Drug: TAB014

INTERVENTIONS:
Drug: TAB014 — TAB014 of 1.25mg(0.05ml)、2.00mg(0.08ml)、2.50mg(0.10ml)
  Other Names: TAB014 monoclonal antibody injection

SUMMARY:
Subjects with secondary wet age-related macular degeneration(AMD) or recurrent subfoveal choroidal neovascularization (CNV) in only one study eye will be enrolled into the study.

DETAILED DESCRIPTION:
The screening period was 28 days. The classification of CNV will be determined by Fundus Fluorescein Angiography ( FFA ) at the study centers. Subjects will receive intravitreal injections of TAB014 Monoclonal Antibody Injection in one eye ( the study eye ). Subjects will only receive single intravitreal dose.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects, 50 years of age or older.
2. Have secondary actively Age-related macular degeneration(wAMD) or recurrent CNV including subfoveal type and extrafoveal type in the only study eye.
3. If have occult CNV or partial classic CNV lesions will be enrolled into the study.
4. The total CNV area(both classic and occult lesion) including lesion area are more than or equal to 50% total lesion areas.
5. The total lesion area is less than or equal to 12 disk area (DA).
6. Volunteer to participate in the study and able to read and understand informed consent and provide written informed consent.

Exclusion Criteria:

1. Prior and concomitant therapy

1. Prior use of verteporfin, external beam radiation therapy or transpupillary thermotherapy(TTT) in 6 months period of the screening.
2. Subjects that have received angiogenesis inhibitors therapy, such as Pegaptanib Sodium, Lucentis, Bevacizumab, Bevacizumab (RETAANE) or protein kinase C inhibitor in either eye are participating in any other research study within the last 6 months before the screening.
3. Subjects that have received other intravitreal injection therapy(Corticosteroids or device implants) in the study eye within the last 6 months before the screening.
4. Subjects that have treated with focal argon laser photocoagulation for macular edema in study eye within the last 6 months before the screening.
5. Subjects that have undergone previous photocoagulation of the retina(extrafoveal areas) in the study eye within the last 3 months before the screening.
6. Subjects with a history of vitreoretinal surgery in the study eye.
7. Subjects that have undergone previous AMD surgery or other surgical interventions.
8. Subjects that have participated in other study of treatment with study drug(except for vitamins and minerals) within the last 3 months before the screening.

2. lesion features:

1. Area of bleeding under the retina 50% total lesion areas or 4 disk area.
2. Subfoveal fibrosis.
3. CNV that be caused by the oter reasons in either eye,such as ocular histoplasmosis syndrome, craniocerebral trauma or pathological myopia.
4. retinal pigment epithelium (RPE) tears. 3. concomitant eye disease:

1) Subjects with ongoing any concomitant eye disease(i.e cataracts or diabetic retinopathy) by the investigator's judgment:

1. Vision loss caused by these diseases to cause interference with medical or operation intervention during 3 months study.
2. Best corrected visual acuity (BCVA) loss at least of 2 lines Snellen equivalents (ETDRS 10 letters) at 3 months, if don't treat the disease.

   2) Subjects who are active endophthalmitis(with micro level or above). 3) Subjects with ongoing internal vitreous hemorrhage. 4) Subjects with Rhegmatogenous retinal detachment or history of macular holes stage 3/4.

   5) Subjects with history of idiopathic uveitis or autoimmune uveitis in either eye 6) Subjects with ongoing infectious conjunctivitis, infectious keratitis, infectious scleral or endophthalmitis in either eye.

   7) Subjects that have undergone previous intraocular surgery (including cataract surgery ) within the last 3 months before the screening.

   8) Subjects who are uncontrolled glaucoma(defined as intraocular pressure [IOP] 30 mmHg, even when treated with anti-glaucoma drugs).

   9) Subjects with history of glaucoma filtration surgery. 4. concomitant system disease:
   1. Subjects of child bearing ages will undergo pregnancy testing.
   2. Subjects with ongoing severe hepatic and renal disease or abnormal liver and kidney function(ALT, Angiotensin sensitivity test (AST) ≥1.5 ULN, Cr, UREA>ULN) at Baseline.
   3. Patients with other disease history,such as uncontrolled diabetics or hypertension, periinfarction within the last 6 months,as well as not suitable for this study per the investigator's judgment.
   4. Subjects with ongoing systemic infection therapy. 5.other:

   <!-- -->

   1. Subjects with history of fluoresceins allergy.
   2. Not get enough quality of fundus photography and fluorescein angiography used by reading and analysing from the reading center.
   3. Unwilling and not be able to return for all study visits

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2018-06-15 (Actual); Primary Completion 2019-02-15 (Estimated); Study Completion 2019-04-30 (Estimated)

PRIMARY OUTCOMES:
Toxicity associated with TAB014 treatment (possibly, probably, or definitively) occurs within 28 days after a single dose of TAB014. | Within 12 weeks after administration
  Describe the impairment of vision by examination.

SECONDARY OUTCOMES:
Dose-limiting toxicity and adverse reaction | Within 12 weeks after administration
  To Assess the dose-limiting toxicity and adverse reaction of TAB014 Monoclonal Antibody Injection.

CONTACTS AND LOCATIONS:
Overall Officials: youxin chen, PHD, Study Director — Peking Union Medical College Hospital of Chinese Academy of Medical Sciences
Locations (1):
- Peking Union Medical College Hospital of Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Schouten JS, La Heij EC, Webers CA, Lundqvist IJ, Hendrikse F. A systematic review on the effect of bevacizumab in exudative age-related macular degeneration. Graefes Arch Clin Exp Ophthalmol. 2009 Jan;247(1):1-11. doi: 10.1007/s00417-008-0952-y. Epub 2008 Oct 9. PMID 18843500
- [Result] Jyothi S, Chowdhury H, Elagouz M, Sivaprasad S. Intravitreal bevacizumab (Avastin) for age-related macular degeneration: a critical analysis of literature. Eye (Lond). 2010 May;24(5):816-24. doi: 10.1038/eye.2009.219. Epub 2009 Aug 14. PMID 19680279
- [Result] Mitchell P. A systematic review of the efficacy and safety outcomes of anti-VEGF agents used for treating neovascular age-related macular degeneration: comparison of ranibizumab and bevacizumab. Curr Med Res Opin. 2011 Jul;27(7):1465-75. doi: 10.1185/03007995.2011.585394. Epub 2011 May 31. PMID 21623685
- [Result] Li J, Zhang H, Sun P, Gu F, Liu ZL. Bevacizumab vs ranibizumab for neovascular age-related macular degeneration in Chinese patients. Int J Ophthalmol. 2013 Apr 18;6(2):169-73. doi: 10.3980/j.issn.2222-3959.2013.02.12. Print 2013. PMID 23638418
- [Result] Kodjikian L, Decullier E, Souied EH, Girmens JF, Durand EE, Chapuis FR, Huot L. Bevacizumab and ranibizumab for neovascular age-related macular degeneration: an updated meta-analysis of randomised clinical trials. Graefes Arch Clin Exp Ophthalmol. 2014 Oct;252(10):1529-37. doi: 10.1007/s00417-014-2764-6. Epub 2014 Aug 22. PMID 25142373
- [Result] Manzano RP, Peyman GA, Khan P, Kivilcim M. Testing intravitreal toxicity of bevacizumab (Avastin). Retina. 2006 Mar;26(3):257-61. doi: 10.1097/00006982-200603000-00001. PMID 16508423
- [Result] Feiner L, Barr EE, Shui YB, Holekamp NM, Brantley MA Jr. Safety of intravitreal injection of bevacizumab in rabbit eyes. Retina. 2006 Oct;26(8):882-8. doi: 10.1097/01.iae.0000230717.85319.f5. PMID 17031287
- [Result] Shahar J, Avery RL, Heilweil G, Barak A, Zemel E, Lewis GP, Johnson PT, Fisher SK, Perlman I, Loewenstein A. Electrophysiologic and retinal penetration studies following intravitreal injection of bevacizumab (Avastin). Retina. 2006 Mar;26(3):262-9. doi: 10.1097/00006982-200603000-00002. PMID 16508424
- [Result] Diabetic Retinopathy Clinical Research Network; Scott IU, Edwards AR, Beck RW, Bressler NM, Chan CK, Elman MJ, Friedman SM, Greven CM, Maturi RK, Pieramici DJ, Shami M, Singerman LJ, Stockdale CR. A phase II randomized clinical trial of intravitreal bevacizumab for diabetic macular edema. Ophthalmology. 2007 Oct;114(10):1860-7. doi: 10.1016/j.ophtha.2007.05.062. Epub 2007 Aug 15. PMID 17698196